CLINICAL TRIAL: NCT05850533
Title: Pilot Feasibility of a Virtual Tai Chi Easy Intervention for Opioid Use Disorder, Anxiety, and Chronic Pain
Brief Title: Tai Chi Easy for Opioid Use Disorder, Anxiety, and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asana Recovery (Other)
Responsible Party: Principal Investigator, Zhanette Coffee, Principal Investigator, Asana Recovery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002492
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Opioid Use Disorder; Chronic Pain; Anxiety
Keywords: Mind-body therapy; Opioid use disorder; Chronic pain; Anxiety; Tai Chi Easy
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi Easy Intervention (Experimental): 8-week/16-session virtual Tai Chi Easy (vTCE) intervention for adults with OUD, anxiety, and chronic pain
  Interventions: Behavioral: Virtual Tai Chi Easy

INTERVENTIONS:
Behavioral: Virtual Tai Chi Easy — Unique to other mind-body therapies, Tai Chi Easy (TCE) is multi-component mind-body therapy including: 1) Gentle movement, 2) Breath practice, 3) Self-massage, and 4) Meditation.

SUMMARY:
A pre-post, single-group, quasi-experimental design will be used to determine the acceptability, feasibility, and appropriateness of a theory-based, 8-week/16-session virtual Tai Chi Easy (vTCE) intervention for adults with OUD, anxiety, and chronic pain. This dissertation has three Aims: 1) Determine the feasibility of an 8-week/16-session, vTCE intervention for adults with OUD, CP, and anxiety; 2) Determine the perceptions of the vTCE intervention participants by conducting a focus group interview post-vTCE; 3) Explore within-subject changes in generalized anxiety, chronic pain intensity, opioid use, opioid cravings, and basic psychological needs post-vTCE.

DETAILED DESCRIPTION:
This study will determine the feasibility of a virtual Tai Chi Easy (vTCE) intervention for adults with opioid use disorder (OUD), chronic pain (CP), and anxiety. OUD is a public health crisis that causes more than 130 deaths daily, costs over $78 billion annually, and disproportionately affects persons with CP and anxiety. CP and anxiety are important contributors to treatment discontinuation and relapse. Interventions that treat the overlapping symptoms of OUD, anxiety, and CP, concurrently, may improve OUD outcomes. Medication Assisted Treatment (MAT) (e.g., Suboxone) is the most common intervention for OUD; yet MAT is underutilized and approximately 50% of people discontinue treatment prematurely or relapse. There is a small but growing body of literature demonstrating that mind-body therapies (e.g., mindfulness, acupuncture, Tai Chi) help improve opioid use, anxiety, pain, self-efficacy, stress, and quality of life. Unique to other mind-body therapies, Tai Chi Easy (TCE) is multi-component mind-body therapy including: 1) Gentle movement, 2) Breath practice, 3) Self-massage, and 4) Meditation. However, the feasibility of vTCE to ameliorate anxiety and CP symptoms among individuals with OUD is not known. This pilot study addresses this gap by examining the feasibility of a vTCE intervention for OUD, CP, and anxiety. A pre-post single-group quasi-experimental design of adults (N=20) with OUD, CP, and anxiety will be recruited from a substance use treatment facility in California. Aim 1, determine the feasibility of an 8-week/16-session, vTCE intervention for adults with OUD, CP, and anxiety using the following benchmarks: a) recruit 20 adults within 2 months, b) at least 75% study retention, c) 80% of data collected, d) at least 80% adherence to vTCE, e) an average rating of 4.0 on intervention acceptability, appropriateness, and feasibility (i.e., three valid 4-item measures, 5-point Likert scale), and f) 0% safety or injury issues during vTCE classes. Aim 2, determine the perceptions of vTCE intervention by conducting a focus group (FG) interview post-vTCE. FG participants (n=8-10) will generate feedback on the vTCE intervention. Aim 3: Explore within-subject changes in generalized anxiety, chronic pain intensity, opioid use, opioid cravings, and basic psychological needs post-vTCE. Exploratory outcome measures will be collected via REDCap at two intervals (pre-vTCE/Week 0) and (post-vTCE/Week 9). Self-report exploratory measures will be collected using the General Anxiety Disorder (GAD-7), chronic pain intensity (GCPS), opioid cravings (OC-VAS scale), and Basic Psychological Needs Satisfaction (BPNS). Changes in opioid use will be collected via urinalysis with a biomarker of opioid use from the outpatient clinic and reported to the principal investigator. A new holistic theoretical framework (Complexity of Opioid Use Disorder Model) will guide this project. Quantitative data will be analyzed using linear regression and Crist and Tanner's five interpretive phases will be used to analyze qualitative data. Results from this study will provide a foundation for conducting a randomized controlled feasibility trial to test vTCE for individuals with OUD, anxiety, and CP.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults 18 years and older
* diagnosed with opioid use disorder and have a coexisting condition (e.g., anxiety AND/OR chronic pain)
* able to read and comprehend 5th grade English and provide informed consent.

Exclusion Criteria:

* subjects cognitively impaired
* active psychosis or current substance use condition requiring a level of care higher than outpatient treatment
* unable to complete study measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Participant Recruitment benchmark | 2 months
  recruit 20 adults within 2 months
Participant Retention benchmark | 8 weeks
  at least 75% study retention, with reasons for attrition collected
Data Collection benchmark | 8 weeks
  80% of data collected, with reasons for missing data or other data collection issues identified
Intervention Adherence benchmark | 8 weeks
  at least 80% adherence to the interventions with class attendance recorded
Intervention Acceptability, Appropriateness and Feasibility | 8 weeks
  an average rating of 4.0 intervention acceptability, appropriateness, and feasibility (i.e., three valid 4-item measures, 5-point Likert scale)
Intervention Safety benchmark | 8 weeks
  0% safety or injury issues during virtual tai chi classes.

SECONDARY OUTCOMES:
perceptions of the virtual tai chi easy | week 9-10 of study
  conducting a virtual focus group interview post-virtual tai chi easy, participants (n=8-10) will generate feedback on the virtual tai chi easy intervention
Generalized anxiety | pre (week 0) and post (week 9)
  General Anxiety Disorder- 7 items (GAD-7)
Chronic pain | pre (week 0) and post (week 9)
  Graded Chronic Pain Scale (GCPS)
Opioid cravings | pre (week 0) and post (week 9)
  opioid cravings (OC-VAS scale)
Basic Psychological Needs | pre (week 0) and post (week 9)
  Basic Psychological Needs Satisfaction (BPNS)
Opioid use | pre (week 0) and post (week 9)
  Changes in opioid use will be collected via a urine drug screen with opioid results (biomarker of opioid use) from the outpatient clinic and reported to PI

CONTACTS AND LOCATIONS:
Locations (1):
- Asana Recovery, Costa Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coffee Z, Badger TA, Taylor-Piliae R, Vanderah TW, Yu CH, Gordon JS. Tai Chi Easy for Opioid Use Disorder: Pilot Feasibility Outcomes and Lessons Learned. J Integr Complement Med. 2025 Nov;31(11):979-986. doi: 10.1177/27683605251360930. Epub 2025 Jul 18. PMID 40681321